CLINICAL TRIAL: NCT07263581
Title: Effect of Hybrid Functional Electrical Stimulation and Augmented Reality-Based Gait Training on Gait Parameters Among Incomplete Spinal Cord Injury Patients
Acronym: FES AR SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Principal Investigator, Prof. Dr. Shoaib Waqas, Professor, Lahore University of Biological and Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UBS24LMSPT012
Record Dates: First submitted 2025-11-16; First posted 2025-12-04 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-11

CONDITIONS: Incomplete Spinal Cord Injury (SCI); ASIA C and D Classification of SCI; Gait Dysfunction
Keywords: Spinal Cord Injury (SCI); Functional Electrical Stimulation (FES); Augmented Reality (AR); Neurorehabilitation; Gait Training; Lower Limb Rehabilitation; T10-L2 Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: This study will use a randomized controlled trial (RCT) with a parallel-group design to compare two gait rehabilitation approaches in individuals with incomplete spinal cord injury (SCI) classified as ASIA C and D. Eligible participants will be randomly assigned to:
  1. Group A (Hybrid Gait Training: Functional Electrical Stimulation + Augmented Reality feedback).
  2. Group B (Conventional Overground Gait Training with mirror/video feedback). Both groups will receive three 30-minute sessions per week for eight weeks under standardized supervision. Pre- and post-intervention assessments will measure gait speed, stride length, cadence, and symmetry using validated tools such as WISCI II, Functional Gait Assessment, and JAKC Observational Gait Analysis. This design enables a direct comparison of traditional versus technology-assisted rehabilitation to inform evidence-based strategies for gait recovery in incomplete SCI.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Hybrid FES-AR Gait Training (Experimental): Hybrid Functional Electrical Stimulation (FES) combined with Augmented Reality (AR) delivers a technology-enhanced gait rehabilitation program for individuals with incomplete spinal cord injury (SCI). FES provides timed electrical activation of lower-limb muscles-including quadriceps, hamstrings, tibialis anterior, and gastrocnemius-synchronized with gait phases to improve muscle recruitment and neuroplasticity. Concurrently, AR overlays real-time visual cues for foot placement, step length, and gait symmetry, supporting motor learning and postural control. Sessions are delivered for 30 minutes, three times per week, over eight weeks, with stimulation parameters individually adjusted for tolerance and functional response.
  Interventions: Device: Functional Electrical Stimulation (FES) and Augmented Reality (AR)
- Active Comparator: Conventional Overground Gait Training (COGT) (Active Comparator): Conventional Overground Gait Training (COGT) is a standard physiotherapy approach used to improve gait performance in individuals with incomplete SCI. Training includes supervised overground walking with visual feedback provided through mirrors or video recordings to support self-correction of gait deviations. Therapy emphasizes step initiation, stride length, cadence, posture, and gait symmetry. Sessions last 30 minutes, three times per week, for eight weeks, conducted under standardized clinical supervision without the use of electrical stimulation or augmented-reality-based visual cues.
  Interventions: Other: Conventional Overground Gait Training (COGT)

INTERVENTIONS:
Device: Functional Electrical Stimulation (FES) and Augmented Reality (AR) — Functional Electrical Stimulation (FES) combined with Augmented Reality (AR) provides an advanced gait rehabilitation approach for individuals with incomplete spinal cord injury (SCI). FES uses controlled electrical currents to activate key lower-limb muscles-including quadriceps, hamstrings, tibialis anterior, and gastrocnemius-synchronized with gait phases via sensor-driven systems, promoting strength, coordination, and neuroplasticity. AR delivers real-time visual cues for step length, foot placement, and gait symmetry, engaging cognitive and neuromuscular pathways to enhance motor learning and spatial awareness. Participants will undergo 30-minute sessions, three times per week, for eight weeks, with stimulation parameters (pulse width 200-400 μs, frequency 30-50 Hz, individualized intensity) tailored to tolerance. This hybrid approach distinguishes itself from conventional training by combining direct neuromuscular activation to optimize gait recovery in incomplete SCI.
  Arms: Experimental: Hybrid FES-AR Gait Training
Other: Conventional Overground Gait Training (COGT) — Conventional Overground Gait Training (COGT) is a standard physiotherapy approach for improving walking ability in individuals with incomplete spinal cord injury (SCI). In this study, participants in the control group will perform walking exercises over ground, guided by a therapist, with visual feedback provided through mirrors or video observation. Training will focus on step initiation, stride length, cadence, and gait symmetry, emphasizing proper posture and safe weight shifting. Sessions will last 30 minutes, three times per week, for eight weeks under standardized clinical supervision. Unlike technology-assisted interventions, COGT relies on voluntary muscle activation and therapist-guided corrections without electrical stimulation or augmented reality cues.
  Arms: Active Comparator: Conventional Overground Gait Training (COGT)

SUMMARY:
The goal of this clinical trial is to determine whether combining Functional Electrical Stimulation (FES) with Augmented Reality (AR)-based gait training can improve walking ability in individuals with incomplete spinal cord injury (SCI). The study aims to identify the most effective rehabilitation approach for enhancing gait performance and functional independence among these patients.

In this study, participants will include:

* Adults aged 18-45 years
* Diagnosed with incomplete spinal cord injury (ASIA Impairment Scale grades C or D)
* Neurological level of injury between T10 and L2
* Medically stable and able to walk with or without assistive devices
* Cognitively intact and capable of providing informed consent

Exclusion Criteria:

* Severe spasticity or contractures in the lower limbs
* Significant pain or joint instability
* Other neurological or musculoskeletal disorders (e.g., stroke, multiple sclerosis)
* Recent lower limb fractures or orthopedic surgeries
* Cardiovascular instability or open skin lesions Two treatment groups will be formed: Group A and Group B.
* Group A will receive Hybrid FES-AR gait training, which combines electrical stimulation of muscles with visual, task-specific feedback provided through augmented reality.
* Group B will receive conventional gait training, which includes standard physiotherapy methods such as strength, balance, and mobility exercises without FES or AR.

Both interventions will be delivered over 12 weeks, with 3 sessions per week, each lasting approximately 40 minutes.

Baseline assessments will be conducted before starting therapy, followed by evaluations at 6 weeks and 12 weeks. The outcome measures will include improvements in gait speed, step length, stride length, cadence, and gait symmetry, using validated clinical tools such as the JAKC Observational Gait Analysis, Walking Index for Spinal Cord Injury II (WISCI II), and the Functional Gait Assessment (FGA).

This study seeks to determine whether the hybrid approach (FES + AR) leads to greater improvement in walking ability compared to traditional gait training. The findings may help guide future rehabilitation strategies and support the integration of technology-based interventions into spinal cord injury management.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) is a debilitating neurological condition characterized by varying degrees of motor and sensory impairment below the level of injury. Individuals with incomplete SCI, particularly those classified as ASIA Impairment Scale (AIS) Grades C and D, retain partial voluntary motor function and therefore demonstrate significant potential for neurological and functional recovery. Despite this capacity, gait abnormalities such as reduced step length, altered cadence, asymmetrical stride, and impaired balance remain common, contributing to limitations in independence, mobility, and quality of life. Enhancing gait performance in this population requires rehabilitation strategies that support neuroplasticity, promote motor relearning, and provide sufficient sensory feedback.

Functional Electrical Stimulation (FES) is an established modality used to generate controlled muscle contractions by stimulating peripheral motor nerves. In individuals with incomplete SCI, FES assists with activating essential lower limb muscle groups; including the quadriceps, hamstrings, and tibialis anterior, to improve joint motion, stabilize limb control, and facilitate gait-related movement patterns. The stimulation also contributes to strengthening neuromuscular pathways necessary for functional ambulation.

Augmented Reality (AR) provides an interactive rehabilitation environment in which digital visual cues are superimposed onto real-world tasks to guide posture, limb placement, cadence, and motor control. AR-based gait training enhances sensorimotor feedback, increases patient engagement, and allows real-time correction of movement deviations. For individuals with incomplete SCI, this feedback facilitates task-specific motor retraining during walking.

The integration of FES with AR-based gait training represents a hybrid approach that simultaneously targets neuromuscular activation and sensorimotor learning. This combined intervention is designed to optimize spatiotemporal gait mechanics by providing synchronized electrical stimulation and visual feedback during repetitive walking tasks. The protocol focuses on muscle groups critical for locomotion at the T10-L2 neurological levels, where preservation of hip flexors, quadriceps, and ankle dorsiflexors plays a central role in functional gait recovery.

This randomized controlled trial will compare the effectiveness of hybrid FES-AR gait training with conventional overground gait training. The intervention follows a structured schedule across an 8-week period, using standardized procedures to ensure consistency across participants. Outcomes will be assessed using validated tools capable of identifying changes in gait quality, symmetry, efficiency, and functional walking capacity. The trial will evaluate improvements in gait speed, step and stride length, cadence, and symmetry to determine whether the hybrid intervention produces superior outcomes relative to traditional physiotherapy approaches.

The findings from this study are expected to contribute to evidence-based advancements in neurorehabilitation by determining whether technology-assisted gait training provides measurable benefits for individuals with incomplete SCI.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with incomplete spinal cord injury (ASIA Impairment Scale C or D)
* Neurological level of injury between T10 and L2
* Aged 18 to 45 years
* Medically stable with no acute complications
* Able to walk with or without assistive devices
* Cognitively intact
* Capable of providing written informed consent
* Stable physical and emotional health
* No history of seizures
* No major urinary or bowel dysfunction

Exclusion Criteria:

* Severe spasticity or contractures in the lower limbs
* Significant pain or joint instability in the lower limbs
* Presence of other neurological (e.g., stroke, multiple sclerosis) or musculoskeletal disorders
* Open skin lesions or ulcerations
* History of fractures or orthopedic surgery in the lower limbs
* Severe cardiovascular conditions

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Change in Step Length (cm) Measured by JAKC Observational Gait Analysis | 8 weeks
  Step length will be measured in centimeters using the JAKC Observational Gait Analysis. The value represents the distance between initial contact of one foot and the subsequent initial contact of the opposite foot. Data will be reported as mean change from baseline to 8 weeks.
Change in Stride Length (cm) Measured by JAKC Observational Gait Analysis | 8 weeks
  Stride length will be quantified in centimeters as the distance between successive initial contacts of the same foot.
Change in Cadence (steps/min) Assessed by JAKC Observational Gait Analysis | 8 weeks
  Cadence will be measured as the number of steps taken per minute during a standardized walking trial.
Change in Gait Symmetry Ratio (unitless) Using JAKC Observational Gait Analysis | 8 weeks
  Gait symmetry will be assessed using a symmetry ratio calculated from left and right step parameters. Lower values indicate greater symmetry.
Walking Index for Spinal Cord Injury II (WISCI II) | 8 weeks
  It evaluates walking function based on the level of physical assistance and use of assistive devices, providing an objective measure of mobility and independence. The scale ranges from 0 to 20, where higher scores indicate greater independence in walking with fewer or no assistive devices. A score of 0 indicates that the person is unable to walk, while a score of 20 indicates that the person can walk independently without any assistive devices.
Functional Gait Assessment (FGA) | 8 weeks
  The Functional Gait Assessment (FGA) is a 10-item, performance-based clinical scale used to assess postural stability and functional mobility during walking. Each item is scored from 0 to 3, resulting in a total score range of 0 to 30, where higher scores indicate better gait performance and balance.
Step Length (centimeters) | 8 weeks
  Step length will be measured using a standardized measuring tape. Participants will walk along a marked walkway, and the distance between consecutive heel strikes of alternating feet will be recorded. The measurement will be taken in centimeters (cm). Higher values indicate improved gait performance.
Stopwatch 10-Meter Walk Test (10MWT) Gait Speed (meters/second) | 8 weeks
  The 10-Meter Walk Test (10MWT) is a standardized measure used to quantify walking speed in individuals with neurological impairments. Participants walk a distance of 10 meters while timing is recorded using a stopwatch. Gait speed is calculated as distance walked (10 meters) divided by time (seconds). The final outcome will be reported as gait speed in meters per second (m/s), with higher values indicating faster walking speed and better functional mobility.

CONTACTS AND LOCATIONS:
Locations (1):
- Lahore University of Biological and Applied sciences, Lahore, Punjab Province, Pakistan